CLINICAL TRIAL: NCT03234777
Title: Evaluating a Knowledge Translation Tool for Parents: A Pilot Randomized Trial
Brief Title: Evaluating a Knowledge Translation Tool for Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Stollery Children's Hospital (Other)
Responsible Party: Principal Investigator, Lauren Albrecht, PhD Student, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Pro00073867
Record Dates: First submitted 2017-07-17; First posted 2017-07-31 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Acute Gastroenteritis; Pediatric ALL; Knowledge Translation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whiteboard animation video (Experimental): 3 minute video on treatment, management of pediatric acute gastroenteritis
  Interventions: Behavioral: Whiteboard animation video
- Regular video (Sham Comparator): 3 minute video on hand washing for infection control
  Interventions: Behavioral: Regular video

INTERVENTIONS:
Behavioral: Whiteboard animation video — Developed via qualitative research with parents of children with acute gastroenteritis.
  Arms: Whiteboard animation video
Behavioral: Regular video — Developed by CDC
  Arms: Regular video

SUMMARY:
Diarrhea and vomiting in children is a common reason to visit the emergency department. There has been a lot of research on how best to treat children with diarrhea and vomiting who visit the emergency department; however, the care children receive varies by healthcare provider and across hospitals. Additionally, there are things parents can do at home to help manage childhood diarrhea and vomiting and potentially avoid a trip to the emergency department. This shows an urgent need for knowledge translation, that is, efforts to align research knowledge and healthcare practice. Actively involving parents in healthcare decisions has the potential to bridge this gap; however, there is little research on the best ways to communicate complex health information to parents of sick kids. In 2013, a national needs assessment was conducted with parents seeking care for their kids in general emergency departments (trekk.ca). This survey showed that 39% of parents looked for information about their child's health prior to coming to the emergency department and that 44% of these parents looked for this information on the internet. This means that the development and evaluation of digital tools to give parents timely and effective child health information has the potential to reduce unnecessary emergency department visits, empower parents in health decision-making, and ultimately improve child health outcomes. In this project, parents will be actively involved in the evaluation of a digital tool, a whiteboard animation video, designed to communicate the best research evidence on the treatment and management of vomiting and diarrhea in children. In this pilot trial, parents in two emergency departments will be randomized to view the video or a sham video, and then provide quantitative and qualitative data on the potential effectiveness of the video, the perceived benefit and value of the knowledge translation intervention for pediatric vomiting and diarrhea, the feasibility of using iPads and an electronic data collection platform to conduct research with this population, the time required to complete data collection, and parents' willingness to participate in future, similar research.

DETAILED DESCRIPTION:
STUDY PURPOSE: The purpose of this pilot randomized trial is to use quantitative and qualitative approaches to achieve the following objectives in the four key pilot trial domains:

1. Scientific domain objectives:

1.a.) To determine the potential effectiveness of a digital knowledge translation tool for parents/caregivers about pediatric acute gastroenteritis (AGE). KT tools are intended to impact end-user experience, including increasing knowledge, influencing healthcare decision making, and use of healthcare resources/services. Comprehension and retention of health information is a key component of the patient experience, a determinant of care instruction follow-through, and the cornerstone of health literacy; therefore, parental knowledge over time will be assessed. In addition to comprehension, educational materials may also influence health decision making; therefore, parental decision regret over time will be assessed to examine this impact in light of the decision to bring their child to the ED for care. Additionally, minimal clinically important differences (MCIDs) will be identified for both knowledge and decision regret outcome measures. Finally, healthcare utilization post-ED visit will be explored as a potential future outcome.

1. b.) To understand the perceived benefit and value of KT tools for parents/caregivers of a child with pediatric AGE, including important components that enhance knowledge and decision making.
2. Process domain objectives:

2.a.) To examine the feasibility of using an electronic, web-based platform for intervention delivery and data collection with this population.

3. Management domain objectives: 3.a.) To assess parent/caregivers' willingness to participate in future, similar research (i.e., full-scale trial).

4. Resource domain objectives: 4.a.) To determine time required for participants to complete data collection forms.

4.b.) To examine the feasibility of using iPads to collect data with parents/caregivers in the ED.

HYPOTHESIS: This pilot trial is not designed to test hypotheses, but rather to gather initial data to justify and inform a future, full-scale trial.

METHODS & DESIGN: This is a parallel-arm, pilot randomized trial.

Recruitment: Consecutive individuals will be approached in the ED waiting room post-triage assessment during data collection recruitment hours (7 days/week, 0700 - 2300). A member of the study team (Research Coordinator, Research Assistant, etc.) will assess inclusion/exclusion criteria and review the information letter. Informed consent will be indicated on iPads as part of the electronic data collection platform.

Interventions: Participants will view the experimental (3 minute, whiteboard animation video on pediatric acute gastroenteritis) and sham control (3 minute, CDC video on hand washing for infection control) interventions on an iPad in the ED waiting room post-triage assessment. Headphones will be provided with the iPad to both groups in the ED to maintain blinding. At the end of data collection in the ED (post-intervention questionnaire 1), participants can select to receive a link to their allocated video via email. Participants from the experimental intervention group that are participating in the qualitative interview will view the whiteboard animation video again at the start of the interview.

Randomization: Blocked randomization with randomly chosen block sizes will be used to ensure equal distribution of participants to intervention and standard care intervention study arms. The blocked randomization sequence will be computer generated. Following sequence generation, the randomization sequence will be entered into a confidential module on the electronic platform. Once the sequence is entered, the randomization module will only be accessible using a confidential password. The randomization sequence will be kept confidential. It will be inaccessible to data collectors/outcome assessors and to the study participants.

After completing the pre-intervention questionnaire, including demographic information and baseline outcome data, on the electronic data collection platform, participants will automatically be randomized to one of the study conditions (i.e., intervention or sham control) based on the randomization sequence. This process will be seamless to participants. After viewing the study condition materials, participants will be automatically directed to the first post-intervention questionnaire.

Blinding: Using an electronic platform for data collection, study group allocation, and intervention viewing will allow participants to access the interventions and provide data independent of the research team. Participants will know they are viewing information on an iPad, but won't know how the content differs between groups because they will be using headphones. Participants and outcome assessors will not be able to determine group allocation and since all data is collected electronically there is no risk of unblinding during data collection, data cleaning and data analysis.

Sample size estimate: Sample size calculations are not required for pilot/feasibility studies as hypothesis testing is not the focus of this research design. Rather, recruitment will take place over a 6-month period and will be evaluated for quantitative and qualitative components as part of the identified process outcome measures. This 6-month period is intended to reflect the seasonal nature of viral gastroenteritis, the most common cause of infection, in temperate climates. Recruitment will take place over the peak infection time of late winter.

Philosophically, qualitative methods do not conduct prospective determinations of a sample size; instead, an adequate sample permits a deep, case oriented analysis that results in a new understanding of experience. In this study, 12-20 interviews with participants are anticipated to see patterns in experiences.

Data collection:

1. Pre-intervention questionnaire (baseline): Participants will complete a pre-intervention questionnaire that includes demographics, knowledge questionnaire, and Decision Regret Scale within the iCare Adventure platform on the iPad.

   **Participants will then be randomized to view the study intervention or the sham control intervention within the electronic platform on the iPad. This process will be seamless for the participants.
2. Post-intervention questionnaire 1 (immediate): After viewing the intervention, participants will complete the knowledge questionnaire and Decision Regret Scale a second time. In addition, participants will complete 2 items assessing their own performance on the knowledge questionnaire and Decision Regret Scale and 1 item regarding the perceived value and benefit of the KT tool. They will also be asked if they would like a video link emailed to them. At the end of this questionnaire, parents will be informed that the post-intervention questionnaire 2 will be emailed to them 4 days after this ED visit for completion at their earliest convenience. Experimental intervention group parents will be asked about participation in a qualitative focus group at this time.
3. Post-intervention questionnaire 2 (4-14 days post-ED visit): Participants will be emailed a secure link on day 4 post-ED discharge to complete the knowledge questionnaire and Decision Regret Scale a third time 2 items assessing their own performance on the knowledge questionnaire and Decision Regret Scale, 3 items related to healthcare utilization, and 3 items related to the perceived value and benefit of the KT tool (if applicable). Reminders to complete post-intervention questionnaire 2 will be sent every third day (day 7, day 10, day 13). The last day for follow-up questionnaire completion will be 14 days post ED visit (10 days after follow-up survey sent to participant). Previous research has demonstrated that 82% of AGE cases are resolved in three days or less and 14 days represents the outer limit for pediatric AGE resolution.
4. Post-intervention semi-structured interview (sub-sample of experimental group): Participants in the experimental group indicating willingness to participate in an in-depth, semi-structured, qualitative interview will be contacted via telephone after completion of post-intervention questionnaire 2. Up to three phone calls will be made to establish interview date/time. Qualitative interviews will take 30-60 minutes to complete and focus on satisfaction with the electronic data collection platform, perceived benefit and value of the KT intervention, and willingness to participate in future, similar research.

Data analysis: All data will be aggregated and analyzed as per the Alberta Health Information Act. Quantitative data will be downloaded from a secure Canadian server to SPSS for data cleaning and analysis. Data cleaning measures may include recoding into categorical variables and comparing and recoding free text responses where appropriate. Descriptive statistics and estimation are the recommended focus of pilot/feasibility trials. Descriptive statistics (e.g., frequencies, measures of variation and spread, etc.) will be calculated to describe the study groups. Analyses will be conducted based on intention-to-treat overall and by site (Stollery, IWK) to identify any differences in the pattern of results.

Qualitative data will be de-identified during verbatim transcription. Prior to analysis, transcripts will be verified by a member of the research team. Qualitative data will be managed and analyzed using NVivo data management software. Qualitative outcomes will be analyzed using thematic analysis by breaking interview text into small units for a detailed, nuanced account of the data. This iterative process will be concurrent to data collection. Thematic analysis will be guided by the hybrid approach of inductive and deductive coding and theme development described by Fereday & Muir-Cochrane (2006). Deductive coding of the interview transcripts will be done first using the semi-structured interview guide as a framework; smaller units of data that emerge inductively will be coded for increased granularity and specificity. To ensure analytic rigor, field notes will be collected during the data collection and analysis process and coded alongside interview data.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or caregiver of a child 16 years old or younger
2. Child is presenting to the ED with vomiting and diarrhea
3. Parent is fluent in English
4. Parent is willing to be contacted for follow-up data collection

Exclusion Criteria:

1. Child has significant chronic gastrointestinal problem or inflammatory bowel disease (i.e., Crohn's Disease, Inflammatory Bowel Disease, Ulcerative Colitis, chronic constipation)
2. Child is taking immunosuppressive therapy or known history of immunodeficiency
3. Child has undergone oral or gastrointestinal surgery within the preceding 7 days
4. Child has had a prior visit to ED for vomiting and diarrhea within the preceding 14 days

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
knowledge questionnaire | 0-14 days (x3)
  Measure 1 (quantitative) of potential effectiveness of the knowledge translation intervention
Decision Regret Scale | 0-14 days (x3)
  Measure 2 (quantitative) of potential effectiveness of the knowledge translation intervention
Health care utilization | 4-14 days
  Measure 3 (quantitative) of potential effectiveness of the knowledge translation intervention
Perceived benefit and value of the knowledge translation intervention for pediatric AGE | 0-14 days (x2) and qualitative interview (experimental group only) after post-intervention 2 questionnaire
  Measure 4 (qualitative) of potential effectiveness of the knowledge translation intervention

SECONDARY OUTCOMES:
Consent rate | 3 months
  Measure 1 (quantitative) Feasibility of using an electronic data collection platform to conduct research with parents/caregivers
Recruitment rate | 3 months
  Measure 2 (quantitative) Feasibility of using an electronic data collection platform to conduct research with parents/caregivers
Data completion rate | 3 months
  Measure 3 (quantitative) Feasibility of using an electronic data collection platform to conduct research with parents/caregivers
Satisfaction with electronic platform | Assessed during qualitative interview (experimental group only) after post-intervention 2 questionnaire
  Measure 4 (qualitative) Feasibility of using an electronic data collection platform to conduct research with parents/caregivers
Time (minutes) to complete study forms | 0-14 days
  Measure 1 (quantitative) time to complete data collection
Time (days) to complete follow-up questionnaire post-discharge | 0-14 days
  Measure 2 (quantitative) time to complete data collection
Number of technical problems with electronic platform during study period | 3 months
  Data quality measure (quantitative)
Number of technical problems as well as lost, stolen or damaged equipment during study period | 3 months
  Measure 1 (quantitative) feasibility of using iPads to collect data in the emergency department with parents/caregivers
Willingness to participate in future similar research | Assessed during qualitative interview after post-intervention 2 questionnaire
  Qualitative measure

CONTACTS AND LOCATIONS:
Overall Officials: Andre Grace, PhD, Principal Investigator — University of Alberta (Supervisor)
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartling L, Elliott SA, Munan M, Scott SD. Web-Based Knowledge Translation Tool About Pediatric Acute Gastroenteritis for Parents: Pilot Randomized Controlled Trial. JMIR Form Res. 2023 May 25;7:e45276. doi: 10.2196/45276. PMID 37227758
- [Derived] Albrecht L, Scott SD, Hartling L. Evaluating a knowledge translation tool for parents about pediatric acute gastroenteritis: a pilot randomized trial. Pilot Feasibility Stud. 2018 Aug 2;4:131. doi: 10.1186/s40814-018-0318-0. eCollection 2018. PMID 30123522